CLINICAL TRIAL: NCT07049289
Title: Randomized Trial for Telemedical Support Versus Standard Treatment to Control Arterial Hypertension
Brief Title: Telemonitoring in Arterial Hypertension
Acronym: REMOTE-Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMOTE-Control-HTN
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Arterial Hypertension; Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients with arterial hypertension randomized to control arm with standard of care without additional interference through study team
- Telemedical treatment (Experimental): Patients randomized to intervention group will receive biweeky telephone calls and adaption of antiyhpertensive medication if needed
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — Patients randomized to intervention group will receive biweeky telephone calls and adaption of antiyhpertensive medication if needed
  Other Names: telemedicine
  Arms: Telemedical treatment

SUMMARY:
Prospective, randomized trial to assess the effects of a telemedical approach of antihypertensive treatment in comparison with standard care.

Total patient number: 60 patients.

* Intervention group: biweekly telephone calls
* Control group: standard of care

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed arterial hypertension with systolic or diastolic blood pressure >140/90 mmHg in standardized office blood pressure measurement
2. Treatment with 1 to ≤4 antihypertensive drug classes
3. Age >18 years
4. Written informed consent

Exclusion Criteria:

1. Pregnancy
2. Participation in other randomized trials
3. Patients under legal supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Time in blood pressure target range from randomization through 6 months | 6 months
  Time in target range of each blood pressure measurement in first 6 months between control and intervention group

SECONDARY OUTCOMES:
Time in target range months 6 to 12 | 6 months (7-12 months)
  Time in target range of each blood pressure measurement between control and intervention group from months 7 to 12
Medication adherence as assessed by blood/urine sampling after 6 and 12 months | 0, 6 and 12 months
  Medication adherence as assessed by blood/urine sampling after 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Centre Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided